CLINICAL TRIAL: NCT02617329
Title: Effects of Extracorporeal Shock Wave Therapy on Shoulder and Neck Pain
Brief Title: Extracorporeal Therapy on Shoulder and Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: KMUH-IRB-20140137
Record Dates: First submitted 2015-11-17; First posted 2015-11-30 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-08

CONDITIONS: Musculoskeletal Disorders
Keywords: Extracorporeal shock wave therapy (ESWT), Neck Pain
MeSH Terms: conditions — Musculoskeletal Diseases; Neck Pain | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cervical flexion (Other): Education have 8 movement home program for flexion, extension, side bending, rotation in neutral position, and rotation in a position of full cervical flexion.
  Interventions: Other: cervical flexion
- Extracorporeal shock wave therapy (ESWT) (Other): The Extracorporeal shock wave therapy (ESWT) was applied on upper trapezius and levator scapulae following parameters 1.5 bar, per intervention 2000 impulse, once a week for three weeks for the experimental group.
  Interventions: Other: Extracorporeal shock wave therapy (ESWT)

INTERVENTIONS:
Other: Extracorporeal shock wave therapy (ESWT) — The Extracorporeal shock wave therapy (ESWT) was applied on upper trapezius and levator scapulae following parameters 1.5 bar, per intervention 2000 impulse, once a week for three weeks for the experimental group
  Arms: Extracorporeal shock wave therapy (ESWT)
Other: cervical flexion — Education have 8 movement home program for flexion, extension, side bending, rotation in neutral position, and rotation in a position of full cervical flexion.
  Arms: cervical flexion

SUMMARY:
The purpose of this research was to investigate the clinical effects on the ESWT treatment of shoulder and neck pain.

DETAILED DESCRIPTION:
Extracorporeal shock wave therapy (ESWT) has been used to treat various musculoskeletal disorders. The beneficial effects of the ESWT included pain alleviation and improvement in local blood circulation. However, few study exploring the effects of the ESWT for subjects with shoulder and neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific shoulder and neck pain
* Ages between 20yr to 45yr
* Shoulder and neck syndrome of upper trapezius and levator scapulae more than 3 months
* No using medicine such as anodyne and muscle relaxants.

Exclusion Criteria:

-

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The change of visual analogue scale (VAS) | Baseline, week 3

CONTACTS AND LOCATIONS:
Overall Officials: Lan Y Guo, Ph.D, Study Chair — Department of Sports Medicine, College of Medicine, Kaohsiung Medical University
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Cote P, Cassidy JD, Carroll L. The Saskatchewan Health and Back Pain Survey. The prevalence of neck pain and related disability in Saskatchewan adults. Spine (Phila Pa 1976) 23 (15): 1689-1698, 1998 Cagnie B, Danneels L, Van Tiggelen D, De Loose V, Cambier D Individual and work related risk factors for neck pain among office workers: a cross sectional study. Eur Spine J 16(5): 679-686, 2007 Lee HY, Yeh WY, Chen CW, Wang JD. psychosocial risk factors of upper extremity musculoskeletal pain in industries of Taiwan: a nationwide study. J Occup Health, 47(4): 311-318, 2005. Sjölander P, Michaelson P, Jaric S Djupsjöbacka M. Sensorimotor disturbances in chronic neck pain--range of motion, peak velocity, smoothness of movement, and repositioning acuity. Man Ther 13(2): 122-131, 2008.